CLINICAL TRIAL: NCT02377427
Title: An Open-label Study to Characterize the Pharmacokinetics and Pharmacodynamics of Mepolizumab Administered Subcutaneously in Children From 6 to 11 Years of Age With Severe Eosinophilic Asthma
Brief Title: Pharmacokinetics and Pharmacodynamics of Mepolizumab Administered Subcutaneously in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 200363; 2014-002666-76 (EudraCT Number)
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Asthma
Keywords: pharmacokinetics; pediatric; Mepolizumab; subcutaneous; eosinophilic asthma; pharmacodynamics
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mepolizumab 40 mg in Part A and B (Experimental): Participants with bodyweight < 40 kg will receive 0.4 milliliter (mL) of reconstituted mepolizumab subcutaneously, in upper arm or thigh.
  Interventions: Drug: Mepolizumab
- Mepolizumab 100 mg in Part A and B (Experimental): Participants with bodyweight >= 40 kg will receive 1.0 mL of reconstituted mepolizumab subcutaneously, in upper arm or thigh.
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab is supplied as 100 mg lyophilised cake in sterile vials for subcutaneous administration in upper arm or thigh. The vial will be reconstituted with sterile water for injection prior to individual use.

SUMMARY:
Mepolizumab is a humanized immunoglobulin G (IgG1) monoclonal antibody (mAb) that exhibits dose proportional and time-independent pharmacokinetics. The study will be conducted in 2 parts. Part A: it will be pharmacokinetic (PK) and pharmacodynamic (PD) study conducted to support the use of mepolizumab in children aged 6 to 11 years with severe eosinophilic asthma and characterize the PK/PD of mepolizumab 40 milligrams (mg) or 100 mg administered subcutaneously depending on participant body weight. Part B: It is a long-term safety / pharmacodynamic phase in which extended treatment for a further 52 weeks will be offered on an optional basis to those subjects eligible for continued treatment. Participants with bodyweight <40 kilogram (kg) will be dosed with mepolizumab 40 mg and participants with body weight >=40 kg will be dosed with mepolizumab 100 mg subcutaneously in upper arm or thigh at Visit 2 (Week 0). Approximately 40 male or female participants aged 6 to 11 years will be screened to achieve approximately 28 eligible participants entering the treatment phase to allow availability of 20 evaluable participants, with a minimum of six participants enrolled in the <40 kg bodyweight group. The total duration of the study will be 22 weeks and will include a run-in period of 1-2 weeks, a treatment period of 12 weeks and a follow-up phase of 8 weeks. A participant will be considered having completed the study if the participant completes all phases of the study including the follow-up phase (Week 20 [visit 8]).

ELIGIBILITY:
Inclusion Criteria:

* Between 6 and 11 years of age inclusive, at the time of screening.
* Diagnosis of severe asthma, defined by the regional asthma guidelines (i.e., National Institute of Health (NIH), Global Initiative for Asthma (GINA), etc.), for at least 12 months prior to Visit 1. If the participant is naïve to the study site, the participant/guardian must self-report a physician diagnosis of asthma and the investigator must confirm by review of medical history with the participant/guardian.
* Eosinophilic airway inflammation that is related to asthma characterized as eosinophilic in nature as indicated by: elevated peripheral blood eosinophil count of >=300 cells per microliter (cells/μL) demonstrated in the past 12 months OR elevated peripheral blood eosinophil count of >=150/μL at visit 1.
* A well-documented requirement for regular treatment with inhaled corticosteroid (>200 μg/day fluticasone propionate drug powder inhaler [DPI] or equivalent daily) in the 12 months prior to Visit 1 with or without maintenance oral corticosteroids (OCS). The ICS dose should represent medium or high dose in children aged 6-11 years of age [GINA, 2015].
* Current treatment with an additional controller medication for at least 3 months or a documented failure in the past 12 months of an additional controller medication for at least 3 successive months. [e.g., long-acting beta-2-agonist (LABA), leukotriene receptor antagonist (LTRA), or theophylline.]
* Forced expiratory volume in one second (FEV1): Persistent airflow obstruction at either Visit 1 or Visit 2 (FEV1 performed prior to first dose of study medication) as indicated by: A pre-bronchodilator FEV1 <110% predicted (Quanjer, 2012) OR FEV1: Forced vital capacity (FVC) ratio <0.8.
* Previously confirmed history of two or more exacerbations requiring treatment with systemic corticosteroids (CS) (intramuscular [IM], intravenous, or oral), in the 12 months prior to visit 1, despite the use of high-dose inhaled corticosteroids (ICS). For participants receiving maintenance CS, the CS treatment for the exacerbations must have been a two-fold increase or greater in the dose.
* No changes in the dose or regimen of baseline ICS and/or additional controller medication during the run-in period.
* Male or female: Females of childbearing potential must commit to consistent and correct use of an acceptable method of contraception for the duration of the trial and for 4 months after the last dose of investigational product. A urine pregnancy test is required of girls of childbearing potential. This test will be performed at the initial screening visit (visit 1) and will be performed at each scheduled study visit prior to the administration of investigational product, and during the early withdrawal and follow-up visits.
* Parent(s)/guardian able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. If applicable, the participant must be able and willing to give assent to take part in the study according to the local requirement.
* For Part B: The subject has completed all study assessments up-to and including Visit 8 and received all 3 doses of investigational product (IP) in Part A
* For Part B: The Principal Investigator (PI) has performed a benefit/risk assessment and this assessment supports continued therapy with mepolizumab.
* The subject's parents (or guardian) have given consent and the subject has given assent for continued treatment

Exclusion Criteria:

* Participants with any history of life threatening asthma (e.g. requiring intubation), immunosuppressive medications intake or immunodeficiency disorder.
* Participants with any medical condition or circumstance making the volunteer unsuitable for participation in the study.
* Significant abnormality of rate, interval, conduction or rhythm in the 12-lead electrocardiogram (ECG), determined by the investigator in conjunction with the age and gender of the child at Visit 1.
* Alanine aminotransferase (ALT), and bilirubin >2x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at Visit 1.
* Positive Hepatitis B Surface Antigen or positive Hepatitis C antibody at Visit 1.
* Parent/guardian has a history of psychiatric disease, intellectual deficiency, substance abuse, or other condition (e.g. inability to read, comprehend and write) which will limit the validity of consent to participate in this study.
* Unwillingness or inability of the participant or parent/guardian to follow the procedures outlined in the protocol.
* Participant who is mentally or legally incapacitated.
* Children who are wards of the state or government.
* A participant will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* Omalizumab: Participants who have received omalizumab within 130 days of Visit 1.
* Other Biologics: Participants who have received any biological (other than omalizumab) to treat inflammatory disease within 5 half-lives of visit 1.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Hypersensitivity: Participants with allergy/intolerance to a monoclonal antibody or biologic.
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-08-25 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (4):
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Madison, Wisconsin
- Japan (3):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Wakayama
- Poland (2):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Tarnów
- United Kingdom (5):
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20057

REFERENCES:
- [Background] Gupta A, Pouliquen I, Austin D, Price RG, Kempsford R, Steinfeld J, Bradford ES, Yancey SW. Subcutaneous mepolizumab in children aged 6 to 11 years with severe eosinophilic asthma. Pediatr Pulmonol. 2019 Dec;54(12):1957-1967. doi: 10.1002/ppul.24508. Epub 2019 Sep 9. PMID 31502421
- [Background] Gupta A, Ikeda M, Geng B, Azmi J, Price RG, Bradford ES, Yancey SW, Steinfeld J. Long-term safety and pharmacodynamics of mepolizumab in children with severe asthma with an eosinophilic phenotype. J Allergy Clin Immunol. 2019 Nov;144(5):1336-1342.e7. doi: 10.1016/j.jaci.2019.08.005. Epub 2019 Aug 16. PMID 31425781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, open-label study to assess the pharmacokinetics (PK) and pharmacodynamics (PD) of mepolizumab 40 or 100 milligrams (mg) subcutaneously administered to participants with severe eosinophilic asthma aged 6-11 years. This study consisted of two parts: Part A and Part B.
Pre-assignment Details: Part A consisted of pre-screening/ screening/ run-in, treatment, and Follow-up. Part B was long-term treatment and Follow-up phase. A total of 44 participants were screened and 36 were enrolled in Part A. Of which, 30 participants continued on treatment in Part B. Study was conducted in 4 countries (Japan, Poland, United Kingdom and United States).
Groups:
- Part A: Mepolizumab 40 mg SC: Participants with bodyweight < 40 kilograms (kg) received 0.4 milliliter (mL) of reconstituted mepolizumab subcutaneously every four weeks, in upper arm or thigh directly from the investigator or designee, under medical supervision. Participant's weight at Week 0 (Visit 2) was considered to select dosage in Part A. Prior to administration, each vial of mepolizumab were reconstituted and swirled gently to enable complete dissolution of the product.
- Part A: Mepolizumab 100 mg SC; Part B: Mepolizumab 100 mg SC: Participants with bodyweight >= 40 kg received 1.0 mL of reconstituted mepolizumab subcutaneously every four weeks, in upper arm or thigh directly from the investigator or designee, under medical supervision. Prior to administration, each vial of mepolizumab were reconstituted and swirled gently to enable complete dissolution of the product. On investigator discretion, injected volume was split between two injection sites and was given as 2 injections of 0.5 mL each if required.
- Part B: Mepolizumab 40 mg SC: Participants with bodyweight < 40 kg received 0.4 mL of reconstituted mepolizumab subcutaneously every four weeks, in upper arm or thigh directly from the investigator or designee, under medical supervision. Prior to administration, each vial of mepolizumab were reconstituted and swirled gently to enable complete dissolution of the product.
- Part B: Mepolizumab 40/100 mg SC: Participants received either 0.4 mL or 1.0 mL of reconstituted mepolizumab depending upon the bodyweight, administered subcutaneously every four weeks, in upper arm or thigh directly from the investigator or designee, under medical supervision. Prior to administration, each vial of mepolizumab were reconstituted and swirled gently to enable complete dissolution of the product. Participants enrolled to <40 kg at Visit 9 (Week 20) were summarized in the 40/100 mg SC group if they had weight >=40 kg at any subsequent visit.
Period: Part A (Up to Week 20)
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Started | 26 | 10 | 0 | 0 | 0
Completed | 22 | 10 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Other: AE of Asthma Exacerbation | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Period: Part B (From Week 20 and up to Week 80)
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Started | 0 | 0 | 16 (Two participants of PartA chose not to continue in PartB;4 shifted to PartB Mepolizumab 40/100mg arm) | 10 | 4
Completed | 0 | 0 | 15 | 10 | 4
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: Mepolizumab 40 mg SC: Participants with bodyweight < 40 kilogram (kg) received 0.4 milliliter (mL) of reconstituted mepolizumab subcutaneously every four weeks, in upper arm or thigh directly from the investigator or designee, under medical supervision. Participant's weight at Week 0 (Visit 2) was considered to select dosage in Part A. Prior to administration, each vial of mepolizumab were reconstituted and swirled gently to enable complete dissolution of the product.
- Total: Total of all reporting groups
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC | Total
Number analyzed (Participants) | 26 | 10 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.0 (1.79) | 10.0 (1.33) | 8.6 (1.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 20 | 5 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Central/South Asian Heritage (Her.) | 1 | 0 | 1
  Japanese Her. | 6 | 1 | 7
  Black or African American (B or Af Am) | 4 | 3 | 7
  White/Caucasian/European Her. | 14 | 6 | 20
  B or Af Am and White-White/Caucasian/European Her. | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Mepolizumab for Part A
Description: PK of mepolizumab was evaluated in participants using Cmax. PK samples were collected at pre-dose on Weeks 4 and 8; and at Weeks 9, 12, 16 and 20 post-dose. Cmax was evaluated by population PK methods and mean and standard error from the final model has been tabulated. Estimates have been presented from the final model centered to mean bodyweights of 27 kg, 50 kg and 70 kg. Note the average bodyweight of 70 kg (mean body weight observed in adults) was not investigated in the study. PK Population included all participants receiving at least one dose of mepolizumab beginning at Visit 2 (Week 0) and having at least one blood sample taken at Visit 3 (Week 4) or thereafter with measurable mepolizumab plasma concentration.
Time Frame: Pre-dose on Weeks 4 and 8; Weeks 9, 12, 16 and 20 post-dose
Population: PK Population
Measure: Mean (Standard Error); unit: Microgram (ug) per mL
Groups:
- Part A: Mepolizumab SC: Participants received mepolizumab 40 or 100 mg SC, depending on participant's bodyweight (40 mg for <40 kg and 100 mg for >=40 kg). Participants received 0.4 mL of reconstituted mepolizumab subcutaneously (for 40 mg dose) or 1.0 mL of reconstituted mepolizumab subcutaneously (for 100 mg dose) every four weeks, in upper arm or thigh directly from the investigator or designee, under medical supervision. Prior to administration, each vial of mepolizumab were reconstituted and swirled gently to enable complete dissolution of the product.
Arm/Group | Part A: Mepolizumab SC
Number analyzed (Participants) | 36
Microgram (ug) per mL
  70 kg | 12.8188 (0.7843)
  50 kg | 16.3412 (0.6364)
  27 kg | 10.1960 (0.3345)

2. Primary Outcome: Area Under Concentration Time Curve to Infinity (AUC [0-inf]) of Mepolizumab for Part A
Description: PK of mepolizumab was evaluated in participants using AUC (0-inf). PK samples were collected at pre-dose on Weeks 4 and 8; and at Weeks 9, 12, 16 and 20 post-dose. AUC (0-inf) was evaluated by population PK methods and mean and standard error from the final model has been tabulated. Estimates have been presented from the final model centered to mean bodyweights of 27 kg, 50 kg and 70 kg. Note the average bodyweight of 70kg (mean body weight observed in adults) was not investigated in the study.
Time Frame: Pre-dose on Weeks 4 and 8; Weeks 9, 12, 16 and 20 post-dose
Population: PK Population
Measure: Mean (Standard Error); unit: Day*ug per mL
Arm/Group | Part A: Mepolizumab SC
Number analyzed (Participants) | 36
Day*ug per mL
  70 kg | 508.23 (41.8036)
  50 kg | 675.20 (35.8980)
  27 kg | 454.39 (15.8876)

3. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) of Mepolizumab During Treatment Period for Part A
Description: PK of mepolizumab was evaluated in participants using t1/2. PK samples were collected at pre-dose on Weeks 4 and 8; and at Weeks 9, 12, 16 and 20 post-dose. T1/2 was evaluated by population PK methods and mean and standard error from the final model has been tabulated. Estimates have been presented from the final model centered to mean bodyweights of 27 kg, 50 kg and 70 kg. Note the average bodyweight of 70kg (mean body weight observed in adults) was not investigated in the study.
Time Frame: Pre-dose on Weeks 4 and 8; Weeks 9, 12, 16 and 20 post-dose
Population: PK Population
Measure: Mean (Standard Error); unit: Days
Arm/Group | Part A: Mepolizumab SC
Number analyzed (Participants) | 36
Days
  70 kg | 20.9583 (1.6520)
  50 kg | 21.8420 (1.0999)
  27 kg | 23.5582 (0.8406)

4. Primary Outcome: Plasma Apparent Clearance (CL/F) of Mepolizumab in Part A
Description: PK of mepolizumab was evaluated in participants using CL/F. PK samples were collected at pre-dose on Weeks 4 and 8; and at Weeks 9, 12, 16 and 20 post-dose. CL was evaluated by population PK methods and mean and standard error from the final model has been tabulated. Estimates have been presented from the final model centered to mean bodyweights of 27 kg, 50 kg and 70 kg. Note the average bodyweight of 70kg (mean body weight observed in adults) was not investigated in the study.
Time Frame: Pre-dose on Weeks 4 and 8; Weeks 9, 12, 16 and 20 post-dose
Population: PK Population
Measure: Mean (Standard Error); unit: Liter (L) per day
Arm/Group | Part A: Mepolizumab SC
Number analyzed (Participants) | 36
Liter (L) per day
  70 kg | 0.1968 (0.01618)
  50 kg | 0.1481 (0.007874)
  27 kg | 0.08803 (0.003078)

5. Primary Outcome: Ratio to Baseline in Absolute Blood Eosinophil Count at Week 12 for Part A
Description: PD of mepolizumab was evaluated in participants using ratio to Baseline in absolute blood eosinophil count. Blood samples were collected at indicated time points. Baseline was defined as the latest value recorded prior to the first dose of mepolizumab. Ratio to Baseline was calculated as post-dose visit value/Baseline value. It was evaluated by Pharmacodynamic Eosinophils (PDe) Population which included all participants receiving at least one dose of mepolizumab beginning at Visit 2 (Week 0) and having at least one Part A blood sample evaluable for blood eosinophil count.
Time Frame: Baseline and Week 12
Population: PDe Population. Only those participants with data available at specific time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of eosinophils in blood
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 22 | 10
Ratio of eosinophils in blood | 0.115 [0.067 to 0.196] | 0.166 [0.087 to 0.318]

6. Primary Outcome: Number of Participants With on Treatment Serious Adverse Events (SAEs) and Non-SAEs for Part B
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinemia are to be categorized as SAE. On-treatment SAEs and non-SAEs are defined as events occurring from the first Part B dose until 28 days following the last Part B dose. Safety Population includes all participants who received at least one dose of mepolizumab beginning at Visit 9.
Time Frame: From Week 20 and up to Week 72
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Number analyzed (Participants) | 16 | 10 | 4
Participants
  Any SAE | 4 | 2 | 1
  Any Non-SAE | 15 | 8 | 4

7. Primary Outcome: Number of Participants With Positive Anti-mepolizumab Binding Antibodies and Neutralizing Antibodies Response for Part B
Description: Blood sample were collected for the determination of anti-mepolizumab binding antibodies and neutralizing antibodies response in Part B at Weeks 44, 68 and 80 prior to study treatment administration. Participant was considered 'Positive' if they had at least one positive post-Baseline anti-drug antibody assay result. All Part B visits (including scheduled and unscheduled) post-Baseline were considered for Any-time Post-Baseline visit derivation. The number of participants with positive anti-mepolizumab binding antibodies and neutralizing antibodies response at Any Time Post Baseline has been presented. The neutralizing antibodies response results only presented for participants with positive anti-drug antibody assay.
Time Frame: From Week 20 and up to Week 80
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Number analyzed (Participants) | 16 | 10 | 4
Participants
  Anti-drug antibody | 0 | 0 | 0
  Neutralizing antibody | 0 | 0 | 0

8. Primary Outcome: Change From Baseline in Sitting Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) for Part B
Description: Sitting blood pressure measurements included SBP and DBP. Measurements were done pre-infusion/injection with the participant sitting, having rested in this position for at least 5 minutes before each reading. The Baseline was defined as the latest value recorded prior to the first dose of mepolizumab. Change from Baseline was defined as value at indicated time point minus Baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 80
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Number analyzed (Participants) | 16 | 10 | 4
Millimeter of mercury
  Sitting DBP, Week 24, n=16,9, 4: number analyzed (Participants) | 16 | 9 | 4
  Sitting DBP, Week 24, n=16,9, 4 | 1.4 (4.22) | -0.9 (6.68) | -0.8 (3.59)
  Sitting DBP, Week 28, n=15,9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 28, n=15,9, 3 | 5.7 (7.13) | 1.6 (5.53) | -4.0 (7.00)
  Sitting DBP, Week 32, n=15 ,9,3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 32, n=15 ,9,3 | 2.3 (5.65) | 3.0 (7.37) | 1.0 (12.49)
  Sitting DBP, Week 36, n=15,8,3: number analyzed (Participants) | 15 | 8 | 3
  Sitting DBP, Week 36, n=15,8,3 | 3.6 (4.73) | 4.9 (11.14) | 1.7 (8.62)
  Sitting DBP, Week 40, n=15,9,3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 40, n=15,9,3 | 2.3 (8.40) | 4.2 (6.82) | -3.7 (4.73)
  Sitting DBP, Week 44, n=15,9 ,3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 44, n=15,9 ,3 | 1.4 (5.62) | 6.2 (7.61) | 3.7 (11.85)
  Sitting DBP, Week 48, n=15,9,3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 48, n=15,9,3 | 3.5 (7.50) | 4.1 (6.15) | 8.7 (3.21)
  Sitting DBP, Week 52, n=15,9,3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 52, n=15,9,3 | 3.5 (7.55) | 1.4 (5.05) | -3.3 (9.61)
  Sitting DBP, Week 56, n=15,9,3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 56, n=15,9,3 | 2.2 (8.47) | 3.6 (7.14) | -0.3 (8.02)
  Sitting DBP, Week 60, n=15,9,3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 60, n=15,9,3 | 0.8 (4.80) | 6.3 (10.77) | -2.3 (8.08)
  Sitting DBP, Week 64, n=15,9,3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 64, n=15,9,3 | 1.7 (3.48) | 3.9 (8.12) | 0.7 (3.06)
  Sitting DBP, Week 68, n=15,9,3: number analyzed (Participants) | 15 | 9 | 3
  Sitting DBP, Week 68, n=15,9,3 | 3.3 (7.08) | 5.3 (7.60) | -2.0 (10.58)
  Sitting DBP, Week 72, n=15,10,4: number analyzed (Participants) | 15 | 10 | 4
  Sitting DBP, Week 72, n=15,10,4 | 2.5 (6.15) | 5.4 (10.42) | 0.5 (10.21)
  Sitting DBP, Week 80, n=12 ,9,2: number analyzed (Participants) | 12 | 9 | 2
  Sitting DBP, Week 80, n=12 ,9,2 | 1.3 (4.60) | 7.4 (7.60) | 0.5 (13.44)
  Sitting SBP, Week 24, n=16, 9, 4: number analyzed (Participants) | 16 | 9 | 4
  Sitting SBP, Week 24, n=16, 9, 4 | 3.3 (7.44) | -2.4 (13.87) | -6.3 (6.95)
  Sitting SBP, Week 28, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 28, n=15, 9, 3 | 9.3 (6.11) | -0.6 (13.47) | -1.0 (5.57)
  Sitting SBP, Week 32, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 32, n=15, 9, 3 | 2.9 (5.59) | 5.6 (12.04) | -2.7 (16.50)
  Sitting SBP, Week 36, n=15, 8, 3: number analyzed (Participants) | 15 | 8 | 3
  Sitting SBP, Week 36, n=15, 8, 3 | 6.3 (9.13) | 9.4 (11.84) | -1.3 (6.43)
  Sitting SBP, Week 40, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 40, n=15, 9, 3 | 5.5 (7.85) | 4.6 (9.74) | -9.3 (12.22)
  Sitting SBP, Week 44, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 44, n=15, 9, 3 | 4.3 (8.50) | 3.8 (8.32) | 3.0 (9.54)
  Sitting SBP, Week 48, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 48, n=15, 9, 3 | 5.5 (8.25) | 4.2 (11.09) | 3.3 (11.68)
  Sitting SBP, Week 52, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 52, n=15, 9, 3 | 7.8 (7.19) | -1.2 (12.04) | -5.0 (17.32)
  Sitting SBP, Week 56, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 56, n=15, 9, 3 | 4.9 (7.81) | 2.1 (10.33) | -9.7 (15.04)
  Sitting SBP, Week 60, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 60, n=15, 9, 3 | 5.7 (8.33) | 2.3 (16.50) | -3.3 (17.62)
  Sitting SBP, Week 64, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 64, n=15, 9, 3 | 5.5 (7.98) | 5.2 (12.09) | -1.3 (15.89)
  Sitting SBP, Week 68, n=15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting SBP, Week 68, n=15, 9, 3 | 8.6 (8.58) | 5.6 (8.75) | 4.3 (10.02)
  Sitting SBP, Week 72, n=15, 10, 4: number analyzed (Participants) | 15 | 10 | 4
  Sitting SBP, Week 72, n=15, 10, 4 | 6.4 (5.79) | 2.7 (10.93) | -3.3 (9.22)
  Sitting SBP, Week 80, n= 12, 9, 2: number analyzed (Participants) | 12 | 9 | 2
  Sitting SBP, Week 80, n= 12, 9, 2 | 3.3 (4.33) | 3.6 (11.82) | 11.5 (0.71)

9. Primary Outcome: Change From Baseline in Sitting Pulse Rate for Part B
Description: Sitting pulse rate measurements were performed pre-infusion/injection with the participant sitting, having rested in this position for at least 5 minutes before each reading. The Baseline was defined as the latest value recorded prior to the first dose of mepolizumab in Part A. Change from Baseline was defined as value at indicated time point minus Baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 80
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Number analyzed (Participants) | 16 | 10 | 4
Beats per minute
  Sitting pulse rate, Week 24, n= 16, 9, 4: number analyzed (Participants) | 16 | 9 | 4
  Sitting pulse rate, Week 24, n= 16, 9, 4 | -3.8 (5.80) | 4.3 (7.50) | 7.0 (16.51)
  Sitting pulse rate, Week 28, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 28, n= 15, 9, 3 | -7.0 (9.02) | 2.7 (4.92) | 1.7 (9.61)
  Sitting pulse rate, Week 32, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 32, n= 15, 9, 3 | -4.8 (9.75) | 4.7 (10.30) | -7.7 (12.01)
  Sitting pulse rate, Week 36, n= 15, 8, 3: number analyzed (Participants) | 15 | 8 | 3
  Sitting pulse rate, Week 36, n= 15, 8, 3 | -0.5 (11.30) | 7.3 (12.28) | 8.0 (7.00)
  Sitting pulse rate, Week 40, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 40, n= 15, 9, 3 | -4.5 (10.84) | 1.7 (14.04) | -4.0 (4.00)
  Sitting pulse rate, Week 44, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 44, n= 15, 9, 3 | -0.7 (13.56) | 3.4 (12.30) | 4.0 (19.31)
  Sitting pulse rate, Week 48, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 48, n= 15, 9, 3 | -2.3 (11.29) | -0.6 (5.64) | -3.0 (8.19)
  Sitting pulse rate, Week 52, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 52, n= 15, 9, 3 | -1.3 (8.41) | -2.1 (9.03) | 11.7 (4.16)
  Sitting pulse rate, Week 56, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 56, n= 15, 9, 3 | -3.8 (8.90) | -1.9 (10.99) | -0.3 (6.66)
  Sitting pulse rate, Week 60, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 60, n= 15, 9, 3 | -3.4 (11.18) | -1.0 (13.86) | 6.3 (14.43)
  Sitting pulse rate, Week 64, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 64, n= 15, 9, 3 | -2.0 (11.16) | 5.0 (11.26) | 8.3 (16.86)
  Sitting pulse rate, Week 68, n= 15, 9, 3: number analyzed (Participants) | 15 | 9 | 3
  Sitting pulse rate, Week 68, n= 15, 9, 3 | -0.9 (8.03) | -2.4 (9.18) | -4.3 (10.97)
  Sitting pulse rate, Week 72, n= 15, 10, 4: number analyzed (Participants) | 15 | 10 | 4
  Sitting pulse rate, Week 72, n= 15, 10, 4 | -5.3 (8.66) | -0.3 (14.21) | -6.0 (6.83)
  Sitting pulse rate, Week 80, n= 11, 9, 2: number analyzed (Participants) | 11 | 9 | 2
  Sitting pulse rate, Week 80, n= 11, 9, 2 | -2.5 (3.33) | 2.1 (7.24) | 13.0 (9.90)

10. Primary Outcome: Number of Participants With Any Time Change From Baseline Relative to Normal Range in Clinical Chemistry Parameters for Part B
Description: Blood samples were collected for analysis of alanine aminotransferase (ALT), alkaline phosphatase (ALP), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT), albumin, protein, bilirubin, creatinine, urate, direct bilirubin, calcium, carbon dioxide (CO2), chloride, glucose, potassium, sodium and urea. Baseline was defined as the latest value recorded prior to the first dose of mepolizumab in Part A. Change from Baseline was defined as value at indicated time point minus Baseline value. All Part B visits (scheduled and unscheduled) post-Baseline were considered for Any-time Post-Baseline visit derivation. If participant had at least one value for categories "To Low" and/or "To High" along with "To Normal or No Change" then participant was counted under "To Low" and/or "To High". If participant had values which belong only to "To Normal or No Change" then participant was counted under "To Normal or No Change" only. Any Time Post-Baseline values have been presented.
Time Frame: Baseline, from Week 20 and up to Week 72
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Number analyzed (Participants) | 16 | 10 | 4
Participants
  ALT; To Low | 0 | 0 | 0
  ALT; To Normal or No Change | 16 | 10 | 4
  ALT; To High | 0 | 0 | 0
  Albumin; To Low | 0 | 0 | 0
  Albumin; To Normal or No Change | 15 | 10 | 4
  Albumin; To High | 1 | 0 | 0
  ALP; To Low | 0 | 0 | 0
  ALP; To Normal or No Change | 16 | 10 | 4
  ALP;To High | 0 | 0 | 0
  AST; To Low | 0 | 0 | 0
  AST; To Normal or No Change | 16 | 10 | 4
  AST; To High | 0 | 0 | 0
  Bilirubin; To Low | 0 | 0 | 0
  Bilirubin; To Normal or No Change | 16 | 9 | 4
  Bilirubin; To High | 0 | 1 | 0
  Calcium; To Low | 0 | 0 | 0
  Calcium; To Normal or No Change | 16 | 7 | 3
  Calcium; To High | 0 | 3 | 1
  CO2; To Low | 6 | 3 | 3
  CO2; To Normal or No Change | 10 | 7 | 1
  CO2; To High | 0 | 0 | 0
  Chloride; To Low | 0 | 0 | 0
  Chloride; To Normal or No Change | 16 | 9 | 4
  Chloride; To High | 0 | 1 | 0
  Creatinine; To Low | 2 | 2 | 0
  Creatinine; To Normal or No Change | 13 | 7 | 4
  Creatinine; To High | 1 | 1 | 0
  Direct Bilirubin; To Low | 0 | 0 | 0
  Direct Bilirubin; To Normal or No Change | 16 | 10 | 4
  Direct Bilirubin; To High | 0 | 0 | 0
  GGT; To Low | 0 | 0 | 0
  GGT; To Normal or No Change | 16 | 10 | 4
  GGT; To High | 0 | 0 | 0
  Glucose; To Low | 1 | 2 | 0
  Glucose; To Normal or No Change | 10 | 4 | 1
  Glucose; To High | 5 | 4 | 3
  Potassium; To Low | 0 | 1 | 0
  Potassium; To Normal or No Change | 16 | 9 | 4
  Potassium; To High | 0 | 0 | 0
  Protein; To Low | 0 | 0 | 0
  Protein; To Normal or No Change | 15 | 10 | 4
  Protein; To High | 1 | 0 | 0
  Sodium; To Low | 0 | 0 | 0
  Sodium; To Normal or No Change | 16 | 10 | 4
  Sodium; To High | 0 | 0 | 0
  Urate; To Low | 0 | 0 | 0
  Urate; To Normal or No Change | 16 | 10 | 4
  Urate; To High | 0 | 0 | 0
  Urea; To Low | 2 | 1 | 1
  Urea; To Normal or No Change | 14 | 9 | 3
  Urea; To High | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Any Time Change From Baseline Relative to Normal Range in Hematology Parameters for Part B
Description: Blood samples were collected for analysis of basophils, eosinophils, leukocyte, monocyte, neutrophils, lymphocyte, platelets, mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), hemoglobin (Hgb), mean corpuscular volume (MCV), erythrocytes, hematocrit, and reticulocytes/erythrocytes (Ret/Ery). Baseline was defined as the latest value recorded prior to first dose of mepolizumab in Part A. Change from Baseline was defined as value at indicated time point minus Baseline value. All Part B visits (scheduled and unscheduled) post-Baseline were considered for Any-time Post-Baseline visit derivation. If participant had at least one value for categories "To Low" and/or "To High" along with "To Normal or No Change" then participant was counted under "To Low" and/or "To High". If participant had values which belong only to "To Normal or No Change" then participant was counted under "To Normal or No Change" only. Any Time Post-Baseline values have been presented.
Time Frame: Baseline, from Week 20 and up to Week 80
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Number analyzed (Participants) | 16 | 10 | 4
Participants
  Basophils; To Low | 0 | 0 | 0
  Basophils; To Normal or No Change | 16 | 10 | 4
  Basophils; To High | 0 | 0 | 0
  Eosinophils;To Low | 11 | 6 | 3
  Eosinophils; To Normal or No Change | 5 | 4 | 0
  Eosinophils;To High | 0 | 0 | 1
  MCH; To Low | 0 | 1 | 0
  MCH; To Normal or No Change | 16 | 9 | 4
  MCH; To High | 0 | 0 | 0
  MCHC;To Low | 0 | 1 | 0
  MCHC; To Normal or No Change | 16 | 9 | 4
  MCHC; To High | 0 | 0 | 0
  MCV; To Low | 0 | 1 | 0
  MCV; To Normal or No Change | 16 | 9 | 4
  MCV; To High | 0 | 0 | 0
  Erythrocytes; To Low | 0 | 0 | 0
  Erythrocytes; To Normal or No Change | 15 | 8 | 3
  Erythrocytes; To High | 1 | 2 | 1
  Hematocrit; To Low | 0 | 2 | 0
  Hematocrit; To Normal or No Change | 16 | 7 | 4
  Hematocrit; To High | 0 | 1 | 0
  Hgb; To Low | 0 | 1 | 0
  Hgb; To Normal or No Change | 16 | 8 | 4
  Hgb; To High | 0 | 1 | 0
  Leukocytes; To Low | 5 | 2 | 1
  Leukocytes; To Normal or No Change | 11 | 7 | 2
  Leukocytes; To High | 0 | 1 | 1
  Lymphocytes; To Low | 0 | 0 | 0
  Lymphocytes; To Normal or No Change | 15 | 9 | 2
  Lymphocytes; To High | 1 | 1 | 2
  Monocytes; To Low | 6 | 2 | 1
  Monocytes; To Normal or No Change | 10 | 8 | 3
  Monocytes; To High | 0 | 0 | 0
  Neutrophils; To Low | 3 | 2 | 2
  Neutrophils; To Normal or No Change | 13 | 5 | 1
  Neutrophils; To High | 0 | 3 | 1
  Platelets; To Low | 0 | 0 | 0
  Platelets; To Normal or No Change | 15 | 10 | 4
  Platelets; To High | 1 | 0 | 0
  Ret/Ery; To Low | 2 | 3 | 1
  Ret/Ery; To Normal or No Change | 12 | 7 | 3
  Ret/Ery;To High | 2 | 0 | 0

12. Primary Outcome: Number of Participants With Abnormal Findings for Urinalysis Parameters in Part B
Description: Urine samples were collected from participants at indicated time points for analysis of urinalysis parameters including Specific gravity and potential of hydrogen (pH) of urine, presence of glucose, protein, blood and ketones in urine by dipstick test. Microscopic examination was performed if blood or protein was abnormal. Only those participants with data available at the specified time points were analyzed.
Time Frame: From Week 20 and up to Week 72
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Number analyzed (Participants) | 10 | 9 | 1
Participants | 7 | 6 | 0

13. Secondary Outcome: Body Weight-adjusted Apparent Clearance of Mepolizumab for Part A
Description: PK samples were collected at pre-dose on Weeks 4 and 8; and at Weeks 9, 12, 16 and 20 post-dose. The body weight-adjusted apparent clearance was compared between adults and participants aged 6 to 11 years old with severe eosinophilic asthma when mepolizumab was administered subcutaneously. Point estimate and 90% confidence interval (CI) for participants aged 6 to 11 years (centered to a mean bodyweight of 70 kg) was compared with the historic adult estimated body-weight adjusted clearance of 0.22 L/day, around which a proposed 80-125% interval was applied i.e. 0.18-0.28 L/day. Assuming an absolute bioavailability of 75% this corresponds to an apparent clearance of 0.29 L/day with the proposed 80% to 125% interval of 0.23 to 0.36 L/day. Note the average bodyweight of 70kg (mean body weight observed in adults) was not observed in the study.
Time Frame: Pre-dose on Weeks 4 and 8; Weeks 9, 12, 16 and 20 post-dose
Population: PK Population
Measure: Mean (90% Confidence Interval); unit: L/day
Arm/Group | Part A: Mepolizumab SC
Number analyzed (Participants) | 36
L/day
  Weight 70kg | 0.1968 [0.1694 to 0.2241]
  Weight 50kg | 0.1481 [0.1348 to 0.1614]
  Weight 27kg | 0.0880 [0.0828 to 0.0932]

14. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-7 (ACQ-7) at Week 12 in Part A
Description: ACQ-7 is a simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or a result of treatment. The ACQ-7 uses a 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 = category for forced expiratory volume in 1 second [FEV1]%). The instrument has a reported high test-retest reproducibility with an intraclass correlation coefficient =0.90. The minimally important change in score is 0.5. Baseline was defined as the latest value recorded prior to the first dose of mepolizumab. Change from Baseline was calculated as score obtained at Week 12 minus Baseline Score. Pharmacodynamic Outcome (PDo) Population included all participants who received at least one dose of mepolizumab beginning at Visit 2 and having at least one Part A assessment of pharmacodynamic outcomes.
Time Frame: Baseline and Week 12
Population: PDo Population. Only those participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 23 | 10
Scores on a scale | -0.414 (1.1354) | 0.082 (1.3432)

15. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire-7 (ACQ-7) at Weeks 4,8,16 and 20 in Part A
Description: ACQ-7 is a simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or a result of treatment. The ACQ-7 uses a 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7=category for FEV1%). The instrument has a reported high test-retest reproducibility with an intraclass correlation coefficient =0.90. The minimally important change in score is 0.5. Baseline was defined as the latest value recorded prior to the first dose of mepolizumab. Change from Baseline was calculated as score obtained at the indicated time point minus Baseline Score. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 4,8,16 and 20
Population: PDo Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 26 | 10
Scores on a scale
  Week 4, n=26, 10 | -0.548 (1.1351) | -0.473 (0.9607)
  Week 8, n=26, 10 | -0.652 (1.2270) | -0.302 (1.2445)
  Week 16, n=23, 10: number analyzed (Participants) | 23 | 10
  Week 16, n=23, 10 | -0.154 (1.2336) | -0.087 (1.2541)
  Week 20, n=24, 10: number analyzed (Participants) | 24 | 10
  Week 20, n=24, 10 | -0.261 (1.2303) | -0.088 (1.0632)

16. Secondary Outcome: Change From Baseline in Childhood Asthma Control Test (C-ACT) at Week 12 for Part A
Description: The C-ACT assesses asthma control in children 4-11 years of age. The C-ACT is a 7-question, 2-part questionnaire, with items 1 to 4 were completed by the child (with assistance from a caregiver, as needed) and items 5 to 7 were completed by the caregiver. A total sum score based upon responses to all items was calculated to provide an overall measure of asthma control. The derived C-ACT score ranges from 0 (maximum impairment) to 27 (no impairment), where higher scores represent a better outcome. Baseline was defined as the latest value recorded prior to the first dose of mepolizumab. Change from Baseline was calculated as score obtained at Week 12 minus Baseline Score.
Time Frame: Baseline and Week 12
Population: PDo Population. Only those participants with data available at specific time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 22 | 10
Scores on a scale | 2.1 (4.45) | -0.3 (5.19)

17. Secondary Outcome: Change From Baseline in C-ACT at Weeks 4,8,16 and 20 in Part A
Description: The C-ACT assesses asthma control in children 4-11 years of age. The C-ACT is a 7-question, 2-part questionnaire, with items 1 to 4 were completed by the child (with assistance from a caregiver, as needed) and items 5 to 7 were completed by the caregiver. A total sum score based upon responses to all items was calculated to provide an overall measure of asthma control. The derived C-ACT score ranges from 0 (maximum impairment) to 27 (no impairment), where higher scores represent a better outcome. Baseline was defined as the latest value recorded prior to the first dose of mepolizumab. Change from Baseline was calculated as score obtained at the indicated time point minus Baseline Score. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 4,8,16 and 20
Population: PDo Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 26 | 10
Scores on a scale
  Week 4, n=26, 10 | 1.8 (4.19) | 2.4 (4.55)
  Week 8, n=26, 10 | 3.0 (5.77) | 1.5 (4.28)
  Week 16, n=23, 10: number analyzed (Participants) | 23 | 10
  Week 16, n=23, 10 | 1.5 (4.62) | -0.7 (5.19)
  Week 20, n=24, 10: number analyzed (Participants) | 24 | 10
  Week 20, n=24, 10 | 1.0 (4.23) | 0.9 (4.28)

18. Secondary Outcome: Number of Participants With on Treatment SAEs and Non-SAEs in Part A
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment or all events of possible drug-induced liver injury with hyperbilirubinemia were categorized as SAE. Participants who received any of the study treatment and had any on-treatment non-SAE or SAE (defined as events occurring from the first dose until 28 days after the last dose of mepolizumab) were considered for analysis.
Time Frame: Up to Week 20
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 26 | 10
Participants
  Any non-SAE | 18 | 6
  Any SAE | 5 | 1

19. Secondary Outcome: Number of Participants With Any Time Change From Baseline Relative to Normal Range in Hematology Parameters in Part A
Description: Blood samples were collected for analysis of basophils, eosinophils, leukocyte, monocyte, neutrophils, lymphocyte, platelet count, MCH, MCHC, Hgb, MCV, erythrocytes, hematocrit, and Ret/Ery. The Baseline was the latest value recorded prior to the first dose of mepolizumab. Change from Baseline was defined as value at indicated time point minus Baseline value. Any time post Baseline = all visits (scheduled and unscheduled) post Baseline was considered for this visit derivation. If participant had at least one value for categories "To Low" and/or "To High" along with "To Normal or No Change" then participant was counted under "To Low" and/or "To High". If participant had values which belong only to "To Normal or No Change" then participant was counted under "To Normal or No Change" only. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). Any Time Post-Baseline values have been presented.
Time Frame: Baseline and up to Week 20
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 26 | 10
Participants
  Basophils; To Low; n=26, 10 | 0 | 0
  Basophils; To Normal or No Change; n=26, 10 | 25 | 10
  Basophils; To High; n=26,10 | 1 | 0
  Eosinophils; To Low; n=26, 10 | 15 | 6
  Eosinophils; To Normal or No Change; n=26, 10 | 10 | 4
  Eosinophils; To High; n=26, 10 | 1 | 0
  Leukocyte; To Low; n=26, 10 | 8 | 2
  Leukocyte; To Normal or No Change; n=26, 10 | 17 | 8
  Leukocyte; To High; n=26, 10 | 1 | 0
  Monocyte; To Low; n=26, 10 | 6 | 3
  Monocyte; To Normal or No Change; n=26, 10 | 19 | 7
  Monocyte; To High; n=26, 10 | 1 | 0
  Neutrophils; To Low; n=26, 10 | 8 | 3
  Neutrophils; To Normal or No Change; n=26, 10 | 16 | 7
  Neutrophils; To High; n=26, 10 | 2 | 0
  Lymphocyte; To Low; n=26, 10 | 4 | 1
  Lymphocyte; To Normal or No Change; n=26, 10 | 20 | 8
  Lymphocyte; To High; n=26, 10 | 2 | 1
  Platelet count; To Low; n=25, 10: number analyzed (Participants) | 25 | 10
  Platelet count; To Low; n=25, 10 | 0 | 1
  Platelet count; To Normal or No Change; n=25, 10: number analyzed (Participants) | 25 | 10
  Platelet count; To Normal or No Change; n=25, 10 | 22 | 9
  Platelet count; To High; n=25, 10: number analyzed (Participants) | 25 | 10
  Platelet count; To High; n=25, 10 | 3 | 0
  MCH; To Low; n=26, 10 | 2 | 0
  MCH;To Normal or No Change; n=26, 10 | 24 | 10
  MCH; To High; n=26, 10 | 0 | 0
  MCHC; To Low n=26, 10 | 1 | 1
  MCHC; To Normal or No Change; n=26, 10 | 25 | 9
  MCHC; To High; n=26, 10 | 0 | 0
  Hgb; To Low; n=26, 10 | 0 | 1
  Hgb; To Normal or No Change; n=26, 10 | 26 | 9
  Hgb; To High; n=26, 10 | 0 | 0
  MCV; To Low; n=26, 10 | 2 | 0
  MCV; To Normal or No Change; n=26, 10 | 24 | 10
  MCV; To High; n=26, 10 | 0 | 0
  Erythrocytes; To Low; n=26, 10 | 0 | 0
  Erythrocytes; To Normal or No Change; n=26, 10 | 21 | 8
  Erythrocytes; To High; n=26, 10 | 5 | 2
  Hematocrit; To Low; n=26, 10 | 0 | 2
  Hematocrit; To Normal or No Change; n=26, 10 | 26 | 8
  Hematocrit; To High; n=26, 10 | 0 | 0
  Reti/Ery; To Low; n=26,10 | 8 | 1
  Reti/Ery;To Normal/No Change;n=26,10 | 15 | 9
  Ret/Ery;To High; n=26,10 | 3 | 0

20. Secondary Outcome: Number of Participants With Any Time Change From Baseline Relative to Normal Range in Clinical Chemistry Parameters in Part A
Description: Blood samples were collected for analysis of ALT, ALP, AST, GGT, albumin, protein, total billirubin, creatinine, direct billirubin, urate, calcium, CO2, chloride, glucose, potassium, sodium and urea. Baseline was defined as the latest value recorded prior to the first dose of mepolizumab. Change from Baseline was defined as value at indicated time point minus Baseline value. Any time post Baseline = all visits (including scheduled and unscheduled) post Baseline was considered for this visit derivation. If participant had at least one value for categories "To Low" and/or "To High" along with "To Normal or No Change" then participant was counted under "To Low" and/or "To High". If participant had values which belong only to "To Normal or No Change" then participant was counted under "To Normal or No Change" only. Any Time Post-Baseline values have been presented.
Time Frame: Baseline and up to Week 20
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 26 | 10
Participants
  ALT; To Low | 0 | 0
  ALT; To Normal or No chang | 26 | 10
  ALT; To High | 0 | 0
  AST;To Low | 0 | 0
  AST;To Normal or No Change | 26 | 10
  AST;To High | 0 | 0
  ALP;To Low | 0 | 0
  ALP;To Normal or No Change | 26 | 10
  ALP;To High | 0 | 0
  GGT;To Low | 0 | 0
  GGT;To Normal or No Change | 26 | 10
  GGT;To High | 0 | 0
  Albumin;To Low | 0 | 0
  Albumin;To Normal or No Change | 22 | 10
  Albumin;To High | 4 | 0
  Protein;To Low | 0 | 0
  Protein;To Normal or No Change | 23 | 10
  Protein;To High | 3 | 0
  Total billirubin;To Low | 0 | 0
  Total billirubin;To Normal or No Change | 26 | 10
  Total billirubin;To High | 0 | 0
  Creatinine;To Low | 4 | 1
  Creatinine;To Normal or No Change | 22 | 9
  Creatinine;To High | 0 | 0
  Direct billirubin;To Low | 0 | 0
  Direct billirubin;To Normal or No Change | 26 | 10
  Direct billirubin;To High | 0 | 0
  Urate;To Low | 1 | 0
  Urate;To Normal or No Change | 25 | 10
  Urate;To High | 0 | 0
  Calcium;To Low | 0 | 0
  Calcium;To Normal or No Change | 22 | 8
  Calcium; To High | 4 | 2
  CO2;To Low | 12 | 3
  CO2;To Normal or No Change | 14 | 7
  CO2;To High | 0 | 0
  Chloride;To Low | 0 | 0
  Chloride;To Normal or No Change | 23 | 9
  Chloride;To High | 3 | 1
  Glucose;To Low | 2 | 0
  Glucose;To Normal or No Change | 17 | 8
  Glucose;To High | 7 | 2
  Potassium;To Low | 0 | 0
  Potassium; To Normal or No Change | 26 | 10
  Potassium;To High | 0 | 0
  Sodium,To Low | 0 | 0
  Sodium;To Normal or No Change | 26 | 10
  Sodium;To High | 0 | 0
  Urea;To Low | 1 | 3
  Urea;To Normal or No Change | 25 | 7
  Urea;To High | 0 | 0

21. Secondary Outcome: Number of Participants With Abnormal Findings for Urinalysis in Part A
Description: Urine samples were collected from participants at indicated time points for analysis of urinalysis parameters including specific gravity and pH of urine, presence of glucose, protein, blood and ketones in urine by dipstick test. Microscopic examination was performed if blood or protein was abnormal. Only those participants with data available at the specified time points were analyzed.
Time Frame: Up to Week 20
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 15 | 7
Participants | 5 | 4

22. Secondary Outcome: Number of Participants With Positive Anti-mepolizumab Binding Antibodies and Neutralizing Antibodies Response in Part A
Description: Blood sample for immunogenicity was collected for anti-mepolizumab binding antibodies and neutralizing antibodies response in Part A at indicated time points prior to study treatment administration. Number of participants with positive anti-mepolizumab binding antibodies and neutralizing antibodies response was summarized. Participant was considered 'Positive' if they had at least one positive post-baseline assay result. Any Time Post Baseline has been presented, which included all visits (including scheduled and unscheduled) post-baseline was considered for this visit derivation. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 16 and 20
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 26 | 10
Participants
  Anti-drug antibody,Any time post-baseline,n=25, 10: number analyzed (Participants) | 25 | 10
  Anti-drug antibody,Any time post-baseline,n=25, 10 | 1 | 1
  Neutralizing antibody,Any time post-baseline,n=1,1: number analyzed (Participants) | 1 | 1
  Neutralizing antibody,Any time post-baseline,n=1,1 | 0 | 0

23. Secondary Outcome: Change From Baseline in Sitting SBP and DBP in Part A
Description: Sitting blood pressure measurements were performed in Part A at indicated time points. Measurements were done pre-infusion/injection with the participant sitting, having rested in this position for at least 5 minutes before each reading. The Baseline was defined as the latest value recorded prior to the first dose of mepolizumab. Change from Baseline was defined as value at indicated time point minus Baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 4, 8, 9, 12, 16 and 20
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 26 | 10
mmHg
  Sitting DBP, Week 4, n=26, 10 | 0.4 (5.72) | 2.1 (3.87)
  Sitting DBP, Week 8, , n=26, 10 | -0.4 (5.45) | 3.4 (7.59)
  Sitting DBP, Week 9, , n=22, 10: number analyzed (Participants) | 22 | 10
  Sitting DBP, Week 9, , n=22, 10 | 1.8 (9.82) | 4.9 (9.13)
  Sitting DBP, Week 12, , n=23, 10: number analyzed (Participants) | 23 | 10
  Sitting DBP, Week 12, , n=23, 10 | 1.5 (8.88) | 0.3 (9.98)
  Sitting DBP, Week 16, , n=23, 10: number analyzed (Participants) | 23 | 10
  Sitting DBP, Week 16, , n=23, 10 | 0.6 (6.99) | 3.9 (7.06)
  Sitting DBP, Week 20, , n=24, 10: number analyzed (Participants) | 24 | 10
  Sitting DBP, Week 20, , n=24, 10 | 0.7 (6.94) | 5.1 (7.03)
  Sitting SBP, Week 4, n=26, 10 | 3.6 (9.92) | -1.9 (8.81)
  Sitting SBP, Week 8, , n=26, 10 | 1.8 (8.65) | -0.2 (6.23)
  Sitting SBP, Week 9, , n=22, 10: number analyzed (Participants) | 22 | 10
  Sitting SBP, Week 9, , n=22, 10 | 2.8 (10.39) | -0.2 (12.04)
  Sitting SBP, Week 12, , n=23, 10: number analyzed (Participants) | 23 | 10
  Sitting SBP, Week 12, , n=23, 10 | 4.3 (9.89) | -2.9 (11.10)
  Sitting SBP, Week 16, , n=23, 10: number analyzed (Participants) | 23 | 10
  Sitting SBP, Week 16, , n=23, 10 | 4.3 (11.53) | -4.6 (9.94)
  Sitting SBP, Week 20, , n=24, 10: number analyzed (Participants) | 24 | 10
  Sitting SBP, Week 20, , n=24, 10 | 5.0 (9.21) | 1.4 (9.91)

24. Secondary Outcome: Change From Baseline in Sitting Pulse Rate in Part A
Description: Sitting pulse rate measurements was performed in Part A at indicated time points. Measurements were done pre-infusion/injection with the participant sitting, having rested in this position for at least 5 minutes before each reading. The Baseline was defined as the latest value recorded prior to the first dose of mepolizumab. Change from Baseline was defined as value at indicated time point minus Baseline value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 4, 8, 9, 12, 16 and 20
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC
Number analyzed (Participants) | 26 | 10
Beats per minute
  Sitting pulse rate, Week 4, n=26, 10 | -4.0 (10.91) | -1.1 (10.56)
  Sitting pulse rate, Week 8, n=26, 10 | -3.2 (9.11) | 1.8 (7.42)
  Sitting pulse rate, Week 9, n=22, 10: number analyzed (Participants) | 22 | 10
  Sitting pulse rate, Week 9, n=22, 10 | -2.9 (8.31) | 2.3 (9.33)
  Sitting pulse rate, Week 12, n=23, 10: number analyzed (Participants) | 23 | 10
  Sitting pulse rate, Week 12, n=23, 10 | -0.8 (8.31) | -0.5 (10.73)
  Sitting pulse rate, Week 16, n=23, 10: number analyzed (Participants) | 23 | 10
  Sitting pulse rate, Week 16, n=23, 10 | -0.6 (7.65) | 3.5 (10.20)
  Sitting pulse rate, Week 20, n=24, 10: number analyzed (Participants) | 24 | 10
  Sitting pulse rate, Week 20, n=24, 10 | -3.9 (13.13) | 1.8 (8.22)

25. Secondary Outcome: Ratio to Baseline in Absolute Blood Eosinophil Count at Weeks 32, 44, 56, 68, 72 and 80 for Part B
Description: Blood samples were collected at the indicated time points for the analysis of eosinophil count. Baseline was defined as the latest value recorded prior to the first dose of mepolizumab in Part A. Ratio to Baseline was calculated as post-dose visit value/Baseline value. The analysis was based on Pharmacodynamic (Blood Eosinophils) (PDe) Population comprised of all participants receiving at least one dose of mepolizumab beginning at Visit 9 and having at least one Part B blood sample taken for blood eosinophil count. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and Weeks 32, 44, 56, 68, 72 and 80
Population: PDe Population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of eosinophils in blood
Arm/Group | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
Number analyzed (Participants) | 16 | 10 | 4
Ratio of eosinophils in blood
  Week 32; n= 15, 10, 4: number analyzed (Participants) | 15 | 10 | 4
  Week 32; n= 15, 10, 4 | 0.161 [0.100 to 0.259] | 0.176 [0.089 to 0.346] | 0.072 [0.021 to 0.247]
  Week 44; n= 15, 10, 4: number analyzed (Participants) | 15 | 10 | 4
  Week 44; n= 15, 10, 4 | 0.157 [0.093 to 0.263] | 0.189 [0.090 to 0.398] | 0.147 [0.012 to 1.781]
  Week 56; n= 15, 10, 4: number analyzed (Participants) | 15 | 10 | 4
  Week 56; n= 15, 10, 4 | 0.149 [0.090 to 0.246] | 0.172 [0.094 to 0.314] | 0.058 [0.015 to 0.220]
  Week 68; n= 14, 10, 4: number analyzed (Participants) | 14 | 10 | 4
  Week 68; n= 14, 10, 4 | 0.133 [0.078 to 0.227] | 0.214 [0.111 to 0.415] | 0.108 [0.009 to 1.271]
  Week 72; n = 15, 10, 4: number analyzed (Participants) | 15 | 10 | 4
  Week 72; n = 15, 10, 4 | 0.148 [0.086 to 0.254] | 0.134 [0.064 to 0.279] | 0.098 [0.073 to 0.130]
  Week 80; n =9, 7, 0: number analyzed (Participants) | 9 | 7 | 0
  Week 80; n =9, 7, 0 | 0.591 [0.245 to 1.429] | 0.647 [0.269 to 1.560] |

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-SAEs were collected in Part A from first Part A dose until 28 days following last Part A dose (up to Week 20) and in Part B from first Part B dose until 28 days following last Part B dose (Up to Week 72).
Description: Serious adverse events (SAEs) and Non-SAEs were collected in members of Safety Population, comprised of all participants who received at least one dose of open label mepolizumab medication.
Arm/Group | Part A: Mepolizumab 40 mg SC | Part A: Mepolizumab 100 mg SC | Part B: Mepolizumab 40 mg SC | Part B: Mepolizumab 100 mg SC | Part B: Mepolizumab 40/100 mg SC
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/10 | 0/16 | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 5/26 | 1/10 | 4/16 | 2/10 | 1/4
Other Adverse Events (participants affected / at risk) | 18/26 | 6/10 | 15/16 | 8/10 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Mepolizumab 40 mg SC (N=26) | Part A: Mepolizumab 100 mg SC (N=10) | Part B: Mepolizumab 40 mg SC (N=16) | Part B: Mepolizumab 100 mg SC (N=10) | Part B: Mepolizumab 40/100 mg SC (N=4)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 2 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Mepolizumab 40 mg SC (N=26) | Part A: Mepolizumab 100 mg SC (N=10) | Part B: Mepolizumab 40 mg SC (N=16) | Part B: Mepolizumab 100 mg SC (N=10) | Part B: Mepolizumab 40/100 mg SC (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Injection site reaction (General disorders) | 5 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 5 | 3 | 1
Croup infectious (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Eczema infected (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 3 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 3 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 2 | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 4 | 3 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Fibrinous bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Adrenal suppression (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eyelid haematoma (Eye disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Adverse food reaction (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 3 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Enuresis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Pnenumonia Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT02377427/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT02377427/SAP_001.pdf